CLINICAL TRIAL: NCT03089476
Title: Hypothesis: Skin Barrier Dysfunction With Altered Expression of Skin Barrier Proteins and Lipids Predicts Early Food Sensitizations in Infants at High Risk of Atopy
Brief Title: Evaluating Skin Barrier Dysfunction in Infants at High Risk of Atopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study will not go forward
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Melissa Robinson, Allergy Fellow, National Jewish Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3083
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Atopic Dermatitis; Eczema; Food Allergy
Keywords: Prevention; Predictors
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Food Hypersensitivity | interventions — MICU1 protein, human; Sensitivity and Specificity

STUDY DESIGN:
Intervention Model Description: Children at high risk of atopy will be followed up to 6 months of age. The investigator will obtain TEWL measurements, skin tape stripping, and questionnaire data each subsequent visit. During the latter 2 visits, skin prick allergy testing will be obtained for milk, egg, and peanut to determine risk of food allergy. Biologic parents will also undergo STS and TEWL measurements on the first visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High Risk Atopic Infants (Other): Infants, who are at high risk of atopy, which will be determined by a validated questionnaire, will be enrolled. Infants will undergo skin tape stripping (STS), transepidermal water loss assessment (TEWL), bacterial swabs, and parental questionnaires at each visit (3 visits total). At the latter 2 visits, infants will also undergo skin prick testing to evaluate for food sensitization.
  Interventions: Other: Evaluating atopy in infants
- Atopic Adults (Other): Parents of infants enrolled in the study will undergo skin tape stripping (STS), transepidermal water loss assessment (TEWL), and complete questionnaires at the first visit.
  Interventions: Other: Evaluating TEWL and STS in adults

INTERVENTIONS:
Other: Evaluating atopy in infants — This study does not have an intervention. There is the evaluation of the predictive value of TEWL and STS in atopic infants at risk of developing eczema and TEWL and STS in parents of infants.
  Other Names: Atopy; Allergies
  Arms: High Risk Atopic Infants
Other: Evaluating TEWL and STS in adults — This study does not have an intervention. There is the evaluation of the predictive value of TEWL and STS in atopic infants at risk of developing eczema and TEWL and STS in parents of infants.
  Other Names: Atopy; Transepidermal water loss; Skin tape stripping
  Arms: Atopic Adults

SUMMARY:
It is hypothesized that food allergy is preceded by atopic dermatitis (AD), due to a disruption of skin barrier which can predispose one to food sensitization through the skin. The central hypothesis is that increased transepidermal water loss (TEWL) assessment and skin tape strip analysis (STS) of lipid and filaggrin breakdown products will be predictive markers for the development of AD. Additionally, the associated changes in TEWL and STS will further improve the identification of infants at risk of early food sensitization, compared to family history alone.

ELIGIBILITY:
Inclusion Criteria:

* Women with physician confirmed pregnancy at a gestational age of ≥ 34 weeks. Infants at high risk for atopy will have one or both parents affected by an allergic disease. Infants at low risk for atopy will have no parent or sibling affected by allergic disease. Biologic parent(s) of infants at high risk of atopy will also be enrolled in the study.

Exclusion Criteria:

* Pregnancy loss or delivery prior to a gestational age of ≥ 34 weeks, a history of substance or alcohol abuse, psychiatric and developmental co-morbidities that would render a subject unable to provide informed consent or perform study-related procedures, AIDS and HIV infection, or a fetus with chromosomal or congenital abnormalities.

Ages: 34 Weeks to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Serial Transepidermal Water Loss (TEWL) | 12 months
  Skin Barrier Assessment measured through serial transepidermal water loss (TEWL) in grams of water/meters-squared/hour

SECONDARY OUTCOMES:
Skin Tape Stripping (STS) and Filaggrin(FLG) breakdown products | Up to 12 months
  Risk of atopic dermatitis as evaluated through FLG breakdown products, lipid composition in the skin, and skin ape strip samples
Skin prick testing to milk, egg, and peanut | 12 months
  Food Allergen Sensitization measured by positive skin prick testing to milk, egg, and peanut measured as positive or negative

CONTACTS AND LOCATIONS:
Overall Officials: Pia Hauk, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walker L, Downe S, Gomez L. Skin care in the well term newborn: two systematic reviews. Birth. 2005 Sep;32(3):224-8. doi: 10.1111/j.0730-7659.2005.00374.x. PMID 16128978
- [Background] Blume-Peytavi U, Hauser M, Stamatas GN, Pathirana D, Garcia Bartels N. Skin care practices for newborns and infants: review of the clinical evidence for best practices. Pediatr Dermatol. 2012 Jan-Feb;29(1):1-14. doi: 10.1111/j.1525-1470.2011.01594.x. Epub 2011 Oct 20. PMID 22011065
- [Background] Elias PM. Lipid abnormalities and lipid-based repair strategies in atopic dermatitis. Biochim Biophys Acta. 2014 Mar;1841(3):323-30. doi: 10.1016/j.bbalip.2013.10.001. Epub 2013 Oct 12. PMID 24128970
- [Background] Mao-Qiang M, Brown BE, Wu-Pong S, Feingold KR, Elias PM. Exogenous nonphysiologic vs physiologic lipids. Divergent mechanisms for correction of permeability barrier dysfunction. Arch Dermatol. 1995 Jul;131(7):809-16. doi: 10.1001/archderm.131.7.809. PMID 7611797
- [Background] Feingold KR, Elias PM. Role of lipids in the formation and maintenance of the cutaneous permeability barrier. Biochim Biophys Acta. 2014 Mar;1841(3):280-94. doi: 10.1016/j.bbalip.2013.11.007. Epub 2013 Nov 18. PMID 24262790
- [Background] Simpson EL, Chalmers JR, Hanifin JM, Thomas KS, Cork MJ, McLean WH, Brown SJ, Chen Z, Chen Y, Williams HC. Emollient enhancement of the skin barrier from birth offers effective atopic dermatitis prevention. J Allergy Clin Immunol. 2014 Oct;134(4):818-23. doi: 10.1016/j.jaci.2014.08.005. PMID 25282563
- [Background] Horimukai K, Morita K, Narita M, Kondo M, Kitazawa H, Nozaki M, Shigematsu Y, Yoshida K, Niizeki H, Motomura K, Sago H, Takimoto T, Inoue E, Kamemura N, Kido H, Hisatsune J, Sugai M, Murota H, Katayama I, Sasaki T, Amagai M, Morita H, Matsuda A, Matsumoto K, Saito H, Ohya Y. Application of moisturizer to neonates prevents development of atopic dermatitis. J Allergy Clin Immunol. 2014 Oct;134(4):824-830.e6. doi: 10.1016/j.jaci.2014.07.060. PMID 25282564
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Kircik LH, Del Rosso JQ. Nonsteroidal treatment of atopic dermatitis in pediatric patients with a ceramide-dominant topical emulsion formulated with an optimized ratio of physiological lipids. J Clin Aesthet Dermatol. 2011 Dec;4(12):25-31. PMID 22191005
- [Background] Kelleher MM, Dunn-Galvin A, Gray C, Murray DM, Kiely M, Kenny L, McLean WHI, Irvine AD, Hourihane JO. Skin barrier impairment at birth predicts food allergy at 2 years of age. J Allergy Clin Immunol. 2016 Apr;137(4):1111-1116.e8. doi: 10.1016/j.jaci.2015.12.1312. PMID 26924469 (Retraction: PMID 33832698 J Allergy Clin Immunol. 2021 Apr;147(4):1527)
- [Background] Peters RL, Allen KJ, Dharmage SC, Tang ML, Koplin JJ, Ponsonby AL, Lowe AJ, Hill D, Gurrin LC; HealthNuts Study. Skin prick test responses and allergen-specific IgE levels as predictors of peanut, egg, and sesame allergy in infants. J Allergy Clin Immunol. 2013 Oct;132(4):874-80. doi: 10.1016/j.jaci.2013.05.038. Epub 2013 Jul 24. PMID 23891354
- [Background] Halken S. Prevention of allergic disease in childhood: clinical and epidemiological aspects of primary and secondary allergy prevention. Pediatr Allergy Immunol. 2004 Jun;15 Suppl 16:4-5, 9-32. doi: 10.1111/j.1399-3038.2004.0148b.x. PMID 15125698
- [Background] Minasyan A, Babajanyan A, Campbell DE, Nanan R. Validation of a Comprehensive Early Childhood Allergy Questionnaire. Pediatr Allergy Immunol. 2015 Sep;26(6):522-9. doi: 10.1111/pai.12415. Epub 2015 Jul 22. PMID 26031325
- [Background] Kelleher MM, O'Carroll M, Gallagher A, Murray DM, Dunn Galvin A, Irvine AD, Hourihane JO. Newborn transepidermal water loss values: a reference dataset. Pediatr Dermatol. 2013 Nov-Dec;30(6):712-6. doi: 10.1111/pde.12106. Epub 2013 Mar 5. PMID 23458265